CLINICAL TRIAL: NCT01921946
Title: A Phase Ⅰ Study to Evaluate the Pharmacokinetic Interactions and Safety Between Fimasartan and Rosuvastatin in Healthy Male Volunteers
Brief Title: To Evaluate the Pharmacokinetic Interactions and Safety Between Fimasartan and Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Collaborators: Kyungpook National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: BR-FMS-CT-116
Record Dates: First submitted 2013-08-08; First posted 2013-08-14 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-08

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A (Other): Fimasartan (7 days) → Fimasartan + Rosuvastatin (7 days)
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin
- Part B (Other): Rosuvastatin (7 days) → Fimasartan + Rosuvastatin (7 days)
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan
Drug: Rosuvastatin

SUMMARY:
A phase Ⅰ study to evaluate the pharmacokinetic interactions and safety between fimasartan and rosuvastatin in healthy male volunteers.

DETAILED DESCRIPTION:
After subjects have signed informed consent voluntarily, they go through screening period for within 21 days.

As period I, subjects of Part A take fimasartan for 7 days and subjects of Part B take rosuvastatin for 7 days.

And then, after wash out for 7 days, as period II, subjects of both Part A and B take fimasartan and rosuvastatin for 7 days.

At each period, subjects of Part A have blood sampling 2nd, 4th, 6th day before medication, 7th day before and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, and 48hour after medication(17 times in each period, 34 times in total).

At each period, subjects of Part B have blood sampling 2nd, 4th, 6th day before medication, 7th day before and 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 8, 12, 24, 48 and 72hour after medication(17 times in each period, 34 times in total).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, aged 20- 55 years at screening.
2. Body weight of ≥ 50 kg and within ± 20% of ideal body weight (IBW)(kg) = {height (cm) - 100} * 0.9
3. No abnormal symptom or sign, based on medical history and physical examination, with no congenital or chronic disease that requires treatment
4. Subject that is considered appropriate for participating in the study by an investigator, based on clinical laboratory test (serology, hematology, clinical chemistry, urinalysis) and ECG, performed within 3 weeks prior to administration of study drug
5. Subjects must be able to listen to and understand the detailed statement of informed consent, and willing to decide to participate in the study, follow the study directions and provide written informed consent

Exclusion Criteria:

1. History of clinically significant hypersensitivity to study drug, any other drug or additives (yellow no.5).
2. History of any illness that may affect the absorption, distribution, metabolism or excretion (hepatobiliary, renal, cardiovascular, endocrine (e.g., hypothyroidism), respiratory, gastrointestinal, hemato-oncology, central nervous system, psychiatric and musculoskeletal system)
3. Hypotension (systolic ≤ 100 mmHg or diastolic ≤ 65 mmHg) or hypertension (systolic ≥ 140 mmHg or diastolic ≥ 90 mmHg), measured at screening
4. Active liver disease, or the levels of ALT(Aspartate Transaminase), AST (Alanin Transaminase) or total bilirubin > 1.5 x the upper limit of normal
5. Creatinine clearance < 80 mL/min (calculated by Cockcroft-Gault formula using serum creatinine)
6. Evidence of hereditary disease, including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
7. History of gastrointestinal disease (i.g., Crohn's disease, active peptic ulcer) or resection operation that may affect the absorption of the study drug (excluding simple appendectomy or herniorrhaphy)
8. History of major injury, surgical operation, or suspected symptom of acute illness (severe infection, trauma, diarrhea or vomiting) within 4 weeks prior to the first administration of study drug
9. History of excessive alcohol abuse (>21 units/week, 1 unit=10g=12.5mL of pure alcohol), or subjects who cannot abstain from drinking for at least 3 days prior to the start of this study and throughout the study period, or excessive smoking (>10 cigarettes/day)
10. Use of any prescribed drugs or herbal remedies within 2 weeks, or use of any over-the-counter medication within 1 week prior to the first administration of study drug, and this will affect this study or the safety of the subjects in the opinion of the investigator
11. Participation in any other study within 3 months prior to the first administration of study drug (The finish time of previous study is the day of the last administration of study drug)
12. Donation of whole blood within 2 months prior to the first administration of study drug, or donation of any blood products within 1 month prior to the first administration of study drug
13. Abnormal diet that may affect absorption, distribution, metabolism and excretion of drugs (*e.g., Grapefruit juice ≥ 1L /day within 7 days prior to administration of study drug)
14. Positive serologic tests (HBsAg, HCV Ab, HIV Ag/Ab, VDRL)
15. Subject that is judged inappropriate for participating in the study by an investigator, based on clinical laboratory test (serology, hematology, clinical chemistry, urinalysis) or any other reason

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
(AUC tau,ss),(Cmax,ss),(Cmin,ss), (Tmax,ss), (t1/2) | 0~72 hour after medication

CONTACTS AND LOCATIONS:
Overall Officials: Young Ran Yoon, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea